CLINICAL TRIAL: NCT04435236
Title: Cervical Erector Spinae Plane Block Versus Interscalene Plexus Block for Pain Relief After Arthroscopic Shoulder Surgery: A Noninferiority Randomized Clinical Study
Brief Title: Cervical Erector Spinae Block Versus Interscalene Block for Shoulder Surgery
Acronym: cESPINas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ilker Ince, Associated Prof. Dr. MD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/142
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Pain, Acute; Opioid Use
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical ESP block group (Active Comparator): Cervical ESP block will be performed as described by Elsharkawy at al. (7).
  Interventions: Procedure: Cervical ESP block
- ISB Block group (Sham Comparator): ISB block will be performed in transverse orientation of the ultrasound probe to visualize the trunks of the brachial plexus between the anterior and middle scalene muscles
  Interventions: Procedure: Cervical ESP block

INTERVENTIONS:
Procedure: Cervical ESP block — Cervical ESP block will be performed as described by Elsharkawy at al. (7). ISB block will be performed in transverse orientation of the ultrasound probe to visualize the trunks of the brachial plexus between the anterior and middle scalene muscles
  Other Names: ISB Block

SUMMARY:
Severe pain after arthroscopic surgery is a common experience for the patients . Different regional anesthetic technique has been applicated for postoperative pain relief . The main goal of regional anesthesia regarding postoperative pain relief is to reduce opioid requirements. The most commonly used approach is Interscalene brachial plexus block (ISB), since it provides effective postoperative analgesia upto 12 hours. Erector spinae plane block (ESPB) has been reported for a variety of indications such as thoracic and abdominal surgery. Recently, a novel description of a T2-3 erector spinae plane (ESP) as an alternative to a BP block for an upper extremity surgical procedure. Following these studies, direct cervical ESP block has been recently performed successfully as both clinical and cadaveric study. The investigators hypothesized that cervical ESP block is as effective as (non-inferior) interscalene brachial plexus block in terms of postoperative analgesia of shoulder surgery. To evaluate the effectiveness of the cervical ESP block, the investigators have designed a randomized study. Primary aim is to evaluate the postoperative opioid consumption. Secondary aim is to evaluate postoperative pain scores by Numeric Rating Scale (0 to 10 point scale).

DETAILED DESCRIPTION:
This study has been designed as a prospective, randomized and single-blind trial. Local ethics committee of Ataturk University has approved the study (B.30.2.ATA.0.01.00/142). After obtaining the patients' written informed consents, we will include a total number of 94 patients (47 patients for each group). The inclusion criteria of the study was considered as age between 18-80, American Society of Anesthesiologists (ASA) status I-III, eligible for regional anesthesia, and unilateral shoulder surgery. The patients who have clotting disorder, contra-indication for regional anesthesia, infection on the injection site, chronic opioid usage, previous same side shoulder surgery, severe Chronic obstructive pulmonary disease (COPD) , diaphragmatic paralysis, BMI 35 or over will be excluded. A computer-generated randomization program will be used to allocate the patient into two groups. Interscalene brachial plexus block group will be named as Group ISB (n=47) and cervical ESP block group will be named as Group cESP (n=47). The assessor of the outcomes will be blinded to the study groups of the patients. Both ISB block and cervical ESP block will be performed under ultrasound guidance in the block room preoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-80
2. ASA I-III
3. Eligible for regional anesthesia
4. Unilateral shoulder surgery

Exclusion Criteria:

1. The patients who have clotting disorder
2. Contra-endication for regional anesthesia
3. Infection on the injection site
4. Chronic opioid usage
5. Previous same side shoulder surgery
6. Severe COPD
7. Diaphragmatic paralysis
8. BMI 35 or over

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours postoperatively
  Iv Patient-controlled analgesia (PCA) with fentanyl (10mcg/cc concentration) will be started for all patients

SECONDARY OUTCOMES:
Postoperative pain scores | 24 hours postoperatively
  A Numeric Rating Scale (0 to 10 point scale) wiil be used for pain evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: İlker İnce, MD, Principal Investigator — Ataturk University Anesthesiology Clinical Research Office

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394
- [Background] Demir U, Ince I, Aksoy M, Dostbil A, Ari MA, Sulak MM, Kose M, Tanios M, Ozmen O. The Effect of Pre-emptive Dexketoprofen Administration on Postoperative Pain Management in Patients with Ultrasound Guided Interscalene Block in Arthroscopic Shoulder Surgery. J Invest Surg. 2021 Jan;34(1):82-88. doi: 10.1080/08941939.2019.1576809. Epub 2019 Apr 9. PMID 30966835
- [Background] Ritchie ED, Tong D, Chung F, Norris AM, Miniaci A, Vairavanathan SD. Suprascapular nerve block for postoperative pain relief in arthroscopic shoulder surgery: a new modality? Anesth Analg. 1997 Jun;84(6):1306-12. doi: 10.1097/00000539-199706000-00024. PMID 9174311
- [Background] Abdallah FW, Wijeysundera DN, Laupacis A, Brull R, Mocon A, Hussain N, Thorpe KE, Chan VWS. Subomohyoid Anterior Suprascapular Block versus Interscalene Block for Arthroscopic Shoulder Surgery: A Multicenter Randomized Trial. Anesthesiology. 2020 Apr;132(4):839-853. doi: 10.1097/ALN.0000000000003132. PMID 32044802
- [Background] Tsui BCH, Mohler D, Caruso TJ, Horn JL. Cervical erector spinae plane block catheter using a thoracic approach: an alternative to brachial plexus blockade for forequarter amputation. Can J Anaesth. 2019 Jan;66(1):119-120. doi: 10.1007/s12630-018-1170-7. Epub 2018 Jun 4. No abstract available. PMID 29868941
- [Background] Hamadnalla H, Elsharkawy H, Shimada T, Maheshwari K, Esa WAS, Tsui BCH. Cervical erector spinae plane block catheter for shoulder disarticulation surgery. Can J Anaesth. 2019 Sep;66(9):1129-1131. doi: 10.1007/s12630-019-01421-9. Epub 2019 Jun 3. No abstract available. PMID 31161549
- [Background] Elsharkawy H, Ince I, Hamadnalla H, Drake RL, Tsui BCH. Cervical erector spinae plane block: a cadaver study. Reg Anesth Pain Med. 2020 Jul;45(7):552-556. doi: 10.1136/rapm-2019-101154. Epub 2020 Apr 21. PMID 32321860